CLINICAL TRIAL: NCT06978777
Title: Effect of Caffeine on Cold-stimulated Brown Adipose Tissue Activity
Acronym: ACROBAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: ACROBAT_V1_1
Record Dates: First submitted 2025-05-02; First posted 2025-05-18 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Brown Adipose Tissue (BAT) Physiology; Cold Exposure
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled cross-over trial in healthy volunteers with random sequence of the two study interventions.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caffeine (Active Comparator): Participants will be administered a single dose of 200mg caffeine orally in study visite A, before exposing to a mild cold stimulus. Resting energy expenditure will be measured before an after administration of caffeine and cold exposure.
  Interventions: Drug: Caffeine (200 mg)
- Placebo (Placebo Comparator): Participants will be administered a single dose of placebo tablet orally in study visite B, before exposing to a mild cold stimulus. Resting energy expenditure will be measured before an after administration of placebo and cold exposure.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Caffeine (200 mg) — single dose of 200mg caffeine orally in study visit A
  Arms: Caffeine
Drug: Placebo — single dose of 1 tablet Placebo in study visit B
  Arms: Placebo

SUMMARY:
The purpose of the study is to asses brown adipose tissue activity after a cold mild stimulus, preceded by 200mg caffeine or placebo administration.

DETAILED DESCRIPTION:
Brown adipose tissue (BAT) activation is typically through beta3-adrenoceptors (beta3-AR), but beta3-alone are less efficacious than cold in activating human BAT. Recent research suggests that adenosine, released during cold exposure, plays a key role in BAT thermogenesis. This study aims to investigate the role of the adenosine A2A receptor (A2AR) in BAT activation through a randomized trial with mild cold exposure and caffeine, a potent A2AR antagonist, to explore new therapeutic strategies for metabolic diseases.

This is a randomized, double-blind, placebo-controlled cross-over trial involving healthy volunteers. The study includes a screening visit and two main study visits (A and B), which will occur in random order.

During the two study visits, resting energy expenditure will be assessed by indirect calorimetry under warm conditions and following mild cold exposure, after administration of either caffeine or placebo. For cold exposure, participants will wear cooling sleeves around the waist, which gradually lower the surface body temperature to 10°C or to the lowest tolerable temperature without inducing shivering.

Additionally, BAT activity will be assessed using 18F-FDG PET/CT, performed 30 minutes after the injection of 75 MBq of 18F-FDG.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5 to 25 kg/m2
* Able to give informed consent as documented by signature
* Moderate caffeine consumption (1 to 3 cups of coffee per day)
* Increase of EE in response to mild cold of ≥ 5% of REE

Exclusion Criteria:

* Known hypersensitivity or allergy to caffeine
* Concomitant medication other than prescription free analgesics (paracetamol and NSAID) and oral contraceptives
* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, cardiac arrhythmia, hypertension, diabetes mellitus, hyper- or hypothyroidism)
* History of depressive disorder or anxiety disorder
* Smoker / habitual tobacco use
* Habitual excessive alcohol use
* Regular consumption of caffeine containing energy drinks
* Weight change of >5% within 3 months prior to inclusion
* Systolic blood pressure >140 mmHg and/or diastolic blood pressure > 95 mmHg.
* Resting heart rate >90 bpm
* Hypersensitivity to cold (e.g. Raynaud syndrome)
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant.
* Enrolment of the investigator, his/her family members, employees, and other dependent persons
* Enrolment into another study using ionizing radiation within the previous 12 months.
* Pregnancy or lactation

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01-21 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
BAT SUVmean | 30 minutes after end of intervention in study visit A and B.
  Description: 18F-FDG uptake into the supra-clavicular brown adipose tissue as determined by 18F-FDG PET-CT after the respective study intervention

SECONDARY OUTCOMES:
BAT SUVmax | 30 minutes after intervention in study visit A and B.
  maximum SUV in supraclavicular adipose tissue (according to BARCIST 1.0) as determined by 18F-FDG PET-CT after the respective study intervention
BAT Volume | 30 minutes after intervention in study visit A and B.
  volume of supraclavicular adipose tissue (according to BARCIST 1.0) as determined by 18F-FDG PET-CT after the respective study intervention.
Cold induced thermogenesis (CIT) | immediately after the intervention (caffeine or placebo)
  rise in energy expenditure above baseline occurring during mild cold exposure in the respective study intervention.
Resting energy expenditure (REE) | immediately after the intervention (caffeine or placebo)
  REE during warm conditions and at the end of cold exposure.
Respiratory exchange ratio (RER): | immediately after the intervention (caffeine or placebo)
  Ratio between carbon dioxide production and oxygen consumption (VCO2/VO2) during the enregy expenditure (EE) measurements.
Skin temperature | immediately after the intervention (caffeine or placebo)
  Changes in skin temperature after mild cold stimulus. It will be measured during the hole study visits during warm condition and after cold stimulation, using wireless temperature sensors (iButton Thermochron) attached to the skin at 11 pre-defined locations
Metabolom and Lipidome profile | immediately after the intervention (caffeine or placebo)
  Plasma metabolome and lipidome profiles.
Caffeine and its metabolites | immediately after the intervention (caffeine or placebo)
  Plasma caffeine and its metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Betz, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Department of Endocrinology, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No